CLINICAL TRIAL: NCT03389828
Title: Qualitative Assessment of the Work-Sleep Relationship
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918021; 18-E-N021
Record Dates: First submitted 2018-01-03; First posted 2018-01-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03-20

CONDITIONS: Sleep Health
Keywords: Focus Group; Health Disparities; Occupational Health; Behaviors; Natural History
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: The study population will consist of approximately 340 focus groups participants.

SUMMARY:
Background:

Sleep that does not last long and is low-quality is tied to a range of serious health issues. These range from obesity to early death. Research has shown that black people who are professionals or managers are more likely to have this kind of sleep than their white counterparts. Black people are also at higher risk than whites for health problems caused by insufficient sleep. Researchers want to learn more about why these differences exist.

Objective:

To study reasons for racial differences in the work-sleep relationship.

Eligibility:

Adults at least 25 years old who:

* Are non-Hispanic black or non-Hispanic white
* Are employed and work 38 or more hours a week
* Live around Raleigh-Durham-Chapel Hill, NC, or Washington, DC

Design:

Participants will be screened with questions. They will give sociodemographic data like job title, annual income level, and gender. They will give their contact information.

Participants will have 1 study visit. They will be in a closed, private conference room. They will join a focus group. The focus groups will be organized by to race, gender, and occupational class.

Participants will give informed consent before the focus group begins.

During the focus group, participants will be asked about their perceptions of health in general, and their typical work day. They will be asked about sleep.

Participants will also fill out a short questionnaire about their job and sleep habits.

Focus groups will be audio recorded. The entire session will last 90 to 120 minutes.

DETAILED DESCRIPTION:
OBJECTIVE:

Prior research has documented racial differences in sleep health by occupational class. While increasing professional responsibility has been associated with shorter sleep duration among non-Hispanic Blacks, increasing professional responsibility appears to be associated with a lower prevalence of short sleep duration among non-Hispanic Whites. The objective of the present study is to investigate reasons for these racial differences in the work-sleep relationship.

STUDY POPULATION:

The study population will range between a minimum of 238 and a maximum of 408 focus groups participants (7-12 members acceptable per focus group). All non-Hispanic black and white adults 25 years of age or older who are currently working at least 38 hours a week will be eligible for inclusion in the study. To mitigate the influence of known cultural differences in sleep behaviors, participation will be limited to English speakers born in the continental United Sates.

DESIGN:

We will conduct 34 demographically homogenous focus groups consisting of 7-12 participants each. Focus groups will be stratified based race, sex, and occupational class, and will be conducted in both North Carolina and the metropolitan DC area. Focus groups will take place in-person and be conducted by a trained facilitator according to a scripted, semi-structured focus group guide. Audio recordings of the focus groups will be transcribed verbatim by a professional transcription service. De-identified transcripts will be reviewed by the study team to identify qualitative themes in the data, which will be coded in an appropriate software program using a double-coding process. Qualitative data analysis will be conducted to identify potential reasons for racial differences in sleep health by occupational class. We will additionally assess variation by other sociodemographic determinants, including sex, education, income, and geographic region.

OUTCOMES MEASURES:

Outcome measures include the themes/patterns regarding potential system-level influences, beliefs, and behaviors that may explain racial differences in the association between occupational class and sleep health.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Non-Hispanic Black or non-Hispanic White
* Female or Male
* 25 years of age or older
* Employed (38 plus hours/week)
* Residing in the area around Raleigh-Durham-Chapel Hill, NC or Silver Spring, MD

EXCLUSION CRITERIA:

* Born outside the continental United States
* Not fluent in English
* Unwilling to provide answers to all screening questions
* Unwilling to provide informed consent

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample - residents from Durham, NC and the surrounding areas as well as residents from Silver Spring, MD and the surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Outcome measures include the themes/patterns regarding potential system-level influences, beliefs, and behaviors that may explain racial differences in the association between occupational class and sleep health. | At the time of the focus group and in more detail during data analysis (coding)
  Data will be analyzed via qualitative coding software to identify themes/patterns in the narratives of participants in focus groups and interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Chandra L Jackson, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (2):
- United States (2):
  - Social and Scientific Systems, Inc., Silver Spring, Maryland
  - Social and Scientific Systems, Inc., Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jackson CL, Redline S, Kawachi I, Williams MA, Hu FB. Racial disparities in short sleep duration by occupation and industry. Am J Epidemiol. 2013 Nov 1;178(9):1442-51. doi: 10.1093/aje/kwt159. Epub 2013 Sep 9. PMID 24018914
- [Background] Luckhaupt SE, Tak S, Calvert GM. The prevalence of short sleep duration by industry and occupation in the National Health Interview Survey. Sleep. 2010 Feb;33(2):149-59. doi: 10.1093/sleep/33.2.149. PMID 20175398
- [Background] Krueger PM, Friedman EM. Sleep duration in the United States: a cross-sectional population-based study. Am J Epidemiol. 2009 May 1;169(9):1052-63. doi: 10.1093/aje/kwp023. Epub 2009 Mar 18. PMID 19299406